CLINICAL TRIAL: NCT07113236
Title: Effectiveness of Two Training Interventions Aimed at Increasing HPV Vaccination Coverage in Four Regions of Colombia
Brief Title: Effectiveness of Interventions for Improving HPV Vaccination Cover
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia, Columbia (Other Government)
Collaborators: Universidad de Cartagena (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C19010300-582
Record Dates: First submitted 2025-06-27; First posted 2025-08-08 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Health Adults; Teenager
Keywords: Human papillomavirus; vaccination; Uterine Cervical Neoplasms; communitarian intervention; Psychosocial Intervention
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: Advisor and counselor for vaccination
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Instructions by Health professional (Experimental): Instructions by health professional
  Interventions: Behavioral: Instructions, advices
- Control (Active Comparator): no instructions
  Interventions: Other: No instructions
- Instructions by teachers (Experimental): Instructions by teachers for vaccination
  Interventions: Behavioral: Instructions, advices

INTERVENTIONS:
Behavioral: Instructions, advices — A first moment: informed conversation and exploration of myths and realities with the aim of exploring the perceptions and attitudes of participating children and adolescents towards the vaccine against HPV-associated cancers through an open and reflective dialogue; a second moment with the presentation of a testimonial video and reflection with the aim of learning from the experiences of others, finding inspiration and motivation in their stories, and feeling connected with other people; and a third moment of 360° feedback with the aim of receiving final information about HPV, HPV-associated cancers, and the importance of vaccination.
  Arms: Instructions by Health professional; Instructions by teachers
Other: No instructions — No instructions for vaccination
  Arms: Control

SUMMARY:
Research Problem and Question: The development of prophylactic vaccines against the human papillomavirus (HPV) marks a major scientific and technological advance in the fight against cervical cancer. However, translating the efficacy of these results into effectiveness in terms of reducing the disease burden in the target population requires the vaccine to be delivered within comprehensive public health programs. HPV vaccination and cervical cancer screening have not been adequately integrated. While studies have evaluated the effectiveness of different educational strategies aimed at increasing HPV vaccination acceptability and coverage, the evidence is still heterogeneous and limited. In this regard, a systematic review emphasizes that the shortcomings of the available research lie in three key aspects: a lack of coordination with the setting where the intervention is delivered, errors in selecting the most appropriate strategy, and inaccuracies in study design and conduct (risk of bias). In Colombia, there are no recent data from the same time period or by regional context that have evaluated the effectiveness of two training interventions aimed at increasing HPV vaccine coverage.

General Objective To evaluate the effectiveness of two training interventions aimed at increasing HPV vaccine coverage in four regions of Colombia.

Materials and methods Pragmatic cluster randomized controlled trial.

The study hypotheses are:

H1: The use of educational interventions does not increase HPV vaccine coverage.

H2: The use of educational interventions increases HPV vaccine coverage.

DETAILED DESCRIPTION:
The inclusion criteria are: public and private educational institutions recognized by the Ministry of National Education, located in municipalities with a reported HPV vaccination coverage rate of less than 25% (using the national 2021 vaccination coverage statistics as a baseline). Parents or guardians, the educational community, and children attending the selected institution will participate. Children must be between the ages of 9 and 17 years old and boys between 9 and 14 years old, in accordance with the guidelines of the Ministry of Health and Social Protection. To estimate the sample size, the method suggested by Campbell and van Brukelen was implemented, which requires the participation of 12 groups of 100 participants (n=1,200). For each municipality, schools will be selected using the official list of educational institutions provided by the Ministry of Education as a sampling framework. Simple random sampling will be used. The randomization and analysis units will be educational institutions randomly assigned in a 1:1:1 ratio to the control or intervention group. All study arms will receive psychosocial training with training from health professionals and teachers from the selected municipalities, defined within the community setting. Within the school-based intervention, the behavioral component will use two strategies implemented with an approach to biopsychosocial models: the health belief model, the theory of planned behavior, social cognitive theory, or the theory of reasoned action. The outcomes to be measured will be: the proportion of participants (boys and girls aged 9-17 years and boys aged 9-14 years, in accordance with the guidelines of the Ministry of Health and Social Protection) exposed to the intervention who receive a dose of vaccine during the first 30 days after the intervention, the degree of acceptability of vaccination, and the effectiveness of the training strategies in increasing HPV vaccination coverage. Statistical analysis will be performed following the "Intent-to-Treat (ITT)" principle. The primary outcome will be assessed between the intervention and control groups using a two-dimensional multilevel model, with participants nested within each educational institution. The model will be adjusted for covariates at the individual level (Level 1: student sex and age) and the educational setting (Level 2: nature of the educational institution, religious education, and geographic area). Data will be analyzed using R software version 4.4.1 (RStudio 2021.09.0).

Expected Impact The development of this project will allow for the design and implementation of a program to improve vaccination coverage with the quadrivalent human papillomavirus (HPV) vaccine in Colombia.

Analysis plan: the primary outcome will be assessed during the first 30 days after administering the intervention, and statistical analysis will be performed following the "Intent-to-Treat (ITT)" principle. The intention-to-treat population is defined as all participants registered for the training intervention, regardless of their compliance. The primary outcome will be measured during the first 30 days after the intervention, emphasizing that receiving at least one dose of HPV vaccination will be considered the outcome of interest. The population exposed to the intervention who has not received the vaccine at the end of the observation period will be followed up by a member of the research group, who will determine, through home visits, whether the non-vaccination was due to lack of consent or assent, or because they were deemed no longer needed (e.g., initiation of sexual activity, teenage pregnancy). If home contact is not feasible, telephone and written (email) communication will be established to determine whether the non-vaccination was a consequence of migration or displacement from the territory. If contact is not feasible, loss to follow-up will be considered. Sensitivity analyses will be performed to assess the robustness of the conclusions based on the percentage of losses to follow-up.

The primary outcome will be assessed in each intervention group and then compared to the control group using a two-dimensional multilevel model, with participants nested within each cluster (educational institution). The model will be adjusted for covariates at the individual level (level 1: student sex and age) and the educational setting (level 2: nature of the educational institution, religious education, and geographic area). Data will be analyzed using R software version 4.4.1 (RStudio 2021.09.0). Descriptive statistics will be applied to the sociodemographic variables. Measures of central tendency and dispersion will be estimated for continuous data, and absolute and relative frequencies will be used for qualitative data. Frequency and distribution will be examined for categorical variables, and normal distribution and homogeneity of variance will be analyzed for continuous variables. For categorical variables, the differences between each intervention group and the control group will be analyzed using Fisher's exact test or Pearson's chi-square test. Continuous variables will be compared between each intervention group and the control group using the Mann-Whitney test or Student's t test, depending on the presence or absence of normal distribution of the data. Multivariate logistic regression will be implemented to adjust the association of interest for the presence of the previously mentioned level one and two covariates.

A Bonferroni correction will be performed for the level of significance. Confidence intervals will be estimated, and the adjusted and unadjusted odds ratios (OR and OR) will be implemented as measures of association. The study protocol must be previously approved by the Ethics Committee of the National Cancer Institute as the executing entity.

ELIGIBILITY:
Inclusion Criteria:

* Public and private educational institutions recognized by the Ministry of National Education, located in municipalities with a reported HPV vaccination coverage rate of less than 25% (using the national vaccination coverage statistics for 2021 as a baseline).
* Each cluster (educational institution) will be made up of parents or guardians, educators, and children enrolled in the institution. Children must be between the ages of 9 and 17 years old and boys between 9 and 14 years old, in accordance with the guidelines of the Ministry of Health and Social Protection.
* Participants must sign informed consent, and the minor must provide informed assent if they are under 14 years old.

Exclusion Criteria:

Children with known hypersensitivity to the active ingredients or any of the excipients of the vaccine, with acute fever, in a state of immunosuppression (e.g., HIV or prolonged use of steroids) or with a coagulation disorder will not be able to be part of the population assigned to the conglomerate.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Acceptability of vaccination | 12 months
  Proportion of participants who would accept vaccination after the training intervention with a score equal to or greater than 4 on a 1 to 5 Likert scale that qualitatively expresses the degree of agreement with HPV vaccination).

CONTACTS AND LOCATIONS:
Overall Officials: Alba Cómbita, Phd, Study Chair — Instituto Nacional de Cancerologia, Columbia; Juliana Rodriguez, Ginecologisth oncologist, Study Chair — Instituto Nacional de Cancerologia, Columbia; Carolina Wiesner, Director, Study Director — Instituto Nacional de Cancerologia, Columbia
Locations (1):
- Instituto Nacional de Cancerología, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No